CLINICAL TRIAL: NCT04122066
Title: The Pulmonary Safety of the New Oral Antihepatitis C Treatment
Brief Title: the Pulmonary Safety of Antihepatitis C Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Omil Saman, Principle investigator, Assiut University
Other Study IDs: safety of antihepatiis C drugs
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- respiratory symptoms reported in studied patients: If Sofosbuvir\Daclatasvir regimen has respiratory side effects or not and the factors increase incidence of respiratory complications
  Interventions: Drug: sofosbuvir \daclatsvir

INTERVENTIONS:
Drug: sofosbuvir \daclatsvir — study the effect of the new oral antihepatitis C drugs on the respiratory system
  Other Names: Sovaldi\Daklinza

SUMMARY:
pulmonary side effects of the new regimen of antihepatitis C

DETAILED DESCRIPTION:
Hepatitis C is a liver disease caused by the hepatitis C virus.The hepatitis C virus is a blood borne virus The most common modes of infection are through exposure to small quantities of blood, through injection drug use, unsafe injection practices, unsafe health care, and the transfusion of unscreened blood and blood products.

An estimated 71 million people have chronic hepatitis C infection. A significant number of those who are chronically infected will develop cirrhosis and or liver cancer. the treatment of hepatitis C virus (HCV) infection has been difficult, particularly in patients with HCV genotype 1. Reasons for the difficulty include the inherent toxicity and limited efficacy of interferon-based therapy, which has been the cornerstone of anti-HCV efforts during the past 2 decades.

Newly available direct-acting antiviral agents (DAAs) have the potential to dramatically improve HCV eradication rates. Despite these new drugs has been characterized by a very low adverse events rate in the published clinical trials Few data are available on pulmonary adverse events based real life studies

ELIGIBILITY:
Inclusion Criteria:

1. HCV RNA positivity .

Exclusion Criteria:

* Child C cirrhosis.
* Clinically manifest liver decompensation :ascites ,encephalopathy, wasting, hepatorenal syndrome.
* Serum albumin less than 2.8 g/dl,total serum bilirubin more than 3 mg/dl ,INR1.7 or more .
* absolute neutrophil counts < 1500\mm3 and\or platelet less than 50,000/mm3.
* HCC except 6 months after concluding intervention aiming at cure with no evidence of activity by dynamic CT or MRI.
* Extrahepatic malignancy except after two years of disease\disease free interval
* In lymphomas and chronic lymphatic leukemia can be initiated immediately after remission based on the treating oncologist's report
* Pregnancy or inability to use effective contraception
* Inadequately controlled diabetes mellitus (HbA1c>9%)
* sever renal impairment in which creatinine clearance < 30 ml\min
* chronic lung diseases .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients diagnosed as HCV positive and eligible for search criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the pulmonary side effect of the new anti HCV medication in our population. | 3 months
  find out the pulmonary side effects of the new anti hepatitis C treatment (sovosbuvir based regimen )

SECONDARY OUTCOMES:
the factors that increase the incidence of pulmonary complications | 3 months
  Identification the factors that increase the incidence of pulmonary complications with the new anti HCV medications

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Mokhtar, Study Director — Assiut University; Nahed Makhlouf, Study Director — Assiut University; Mostafa kamal, Study Director — Assiut University